CLINICAL TRIAL: NCT05078801
Title: Comparison of Efficacy and Safety of Endoscopic Biliary Drainage and Percutaneous Transhepatic Biliary Drainage for the Management of Perihilar Malignant Biliary Obstruction: a Monocentric Retrospective Study
Brief Title: Endoscopic Versus Radiologic Biliary Drainage for Perihilar Malignant Obstruction
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PI073
Record Dates: First submitted 2021-08-05; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-07

CONDITIONS: Perihilar Cholangiocarcinoma; Jaundice, Obstructive
Keywords: ERCP; EUS-guided biliary drainage; Percutaneous transhepatic biliary drainage; hilar obstruction
MeSH Terms: conditions — Klatskin Tumor; Jaundice, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endoscopic drainage: All patients with perihilar malignant biliary obstruction treated with endoscopic drainage. This drainage can be multimodal using endoscopic retrograde cholangiopancreatography (ERCP) or endoscopic ultrasound (EUS)-guided biliary drainage.
  Interventions: Procedure: Endoscopic drainage
- Radiologic percutaneous drainage: All patients with perihilar malignant biliary obstruction treated with percutaneous drainage
  Interventions: Procedure: Percutaneous transhepatic biliary drainage

INTERVENTIONS:
Procedure: Endoscopic drainage — ERCP and/or EUS-guided biliary drainage
  Groups: Endoscopic drainage
Procedure: Percutaneous transhepatic biliary drainage — US or CT-guided percutaneous drainage
  Groups: Radiologic percutaneous drainage

SUMMARY:
This retrospective monocentric study aims at comparing multimodality endoscopic biliary drainage versus percutaneous radiologic biliary drainage in case of perihilar malignant obstruction.

Data from patients admitted in the Nancy University Hospital, France, between january 2016 and march 2022 with jaundice and perihilar obstruction will be retrospectively collected.

ELIGIBILITY:
Inclusion Criteria:

* hospitalization between january 2006 and march 2022
* perihilar obstruction
* indication of biliary drainage

Exclusion Criteria:

* distal biliary obstruction
* perihilar obstruction without indication of biliary drainage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all adults patients hospitalized in Nancy University Hospital with perihilar biliary malignant obstruction who underwent either endoscopic or percutaneous approach for biliary drainage.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Bilirubin serum level | 7 days
  Diminution of 20% of more on day 7 of the bilirubin serum level

SECONDARY OUTCOMES:
Complications | 16 years
  complication-free survival
number of procedures | 16 years
  total number of procedures, including all endoscopic and radiological interventions
bilirubin serum level on day 30 and on day 90 | 90 days
median survival in months | 16 years
  median survival in month in each group
number of unplanned hospital admissions | 16 years
  total number of unplanned hospital admissions (for unplanned biliary drainage, cholangitis or other complications...)

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy Hospital Center, Nancy, France